CLINICAL TRIAL: NCT06009653
Title: Effect of Tirzepatide Plus Intensive Lifestyle Therapy on Body Weight and Metabolic Health in Latinos With Obesity
Brief Title: Effects of Tirzepatide Plus Intensive Lifestyle Therapy on Body Weight and Metabolic Health in Latinos With Obesity
Acronym: TRZ
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was discontinued prematurely for administrative reasons
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202209182; P50MD017344 (NIH)
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Metabolic Disease
Keywords: Latinos; Obesity; Plant-forward diet; Tirzepatide
MeSH Terms: conditions — Obesity; Metabolic Diseases | interventions — Standard of Care; Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Standard Care (Active Comparator): In this arm, participants will receive the standard care intervention from community health workers.
  Interventions: Behavioral: Standard Care
- Intensive lifestyle intervention plus placebo (Experimental): In this arm, participants will receive a culturally-tailored dietary and behavioral intensive lifestyle intervention from community health workers, and will receive placebo subcutaneous injections weekly during the 52-week intervention.
  Interventions: Behavioral: Culturally-tailored dietary and behavioral intensive lifestyle intervention; Drug: Placebo
- Intensive lifestyle intervention plus tirzepatide (Experimental): In this arm, participants will receive the behavioral plant-based intervention from community health workers, and will receive subcutaneous injections of tirzepatide weekly during the 52-week intervention
  Interventions: Behavioral: Culturally-tailored dietary and behavioral intensive lifestyle intervention; Drug: Tirzepatide

INTERVENTIONS:
Behavioral: Standard Care — Participants will meet with community health workers to receive general health information through individual check-ins.
  Arms: Standard Care
Behavioral: Culturally-tailored dietary and behavioral intensive lifestyle intervention — Participants will meet with community health workers to receive information focused on healthy eating while still adhering to a culturally-tailored plant-forward diet.
  Arms: Intensive lifestyle intervention plus placebo; Intensive lifestyle intervention plus tirzepatide
Drug: Placebo — Participants will receive placebo subcutaneous injections.
  Arms: Intensive lifestyle intervention plus placebo
Drug: Tirzepatide — Participants will receive subcutaneous injections of tirzepatide that gradually increase up to 15 mg per week.
  Arms: Intensive lifestyle intervention plus tirzepatide

SUMMARY:
The purpose of this study is to conduct a three-arm 52-week, randomized controlled trial with double blind treatment to evaluate the effects of a drug called tirzepatide in combination with an innovative, culturally-appropriate, intensive lifestyle intervention (ILI) delivered by community health workers (CHWs) in Latino adults with obesity. Participants will be randomized to 1) standard care (SC, n=25); 2) culturally-tailored dietary and behavioral intensive lifestyle intervention (ILI, n=25) provided by CHWs plus placebo; or 3) ILI plus tirzepatide (ILI-TRZ) for 52 weeks to evaluate the intervention's effect on: i) weight loss; ii) clinical efficacy (change in body fat mass, liver fat, intra-abdominal fat mass and intrahepatic triglyceride content, oral glucose tolerance, glycemic control, insulin sensitivity and b-cell function, plasma lipids, blood pressure, sleep duration, quality and behaviors, physical performance scores); iii) adherence and fidelity to the intervention (adherence to the intervention and barriers to long term adherence, quality-of-life, fidelity of the implementation by CHWs, CHW's and study participants' acceptability and satisfaction with the intervention and eating behaviors. Placebo or tirzepatide will be injected subcutaneously in the abdomen or thigh once a week for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Hispanic and/or Latino heritage
* Body Mass Index (BMI) 30-42 kg/m²
* HbA1c ≤ 6.4%

Exclusion Criteria:

* Previous diagnosis of diabetes or fasting glucose ≥ 126 mg/dl or 2 hr oral glucose tolerance test plasma glucose ≥ 200 mg/dl
* Unstable weight (≥4% during the last 2 months prior to study enrollment)
* CPAP treatment for obstructive sleep apnea
* Severe cardiovascular disease within the 6 months prior to study enrollment
* Severe organ system dysfunction
* Known clinically significant gastric emptying abnormality
* History of chronic or acute pancreatitis
* Thyroid-stimulating hormone (TSH) >1.5X the upper limit of normal
* Medical conditions that cause obesity
* History of significantly active or unstable Major Depressive Disorder or other severe psychiatric disorder within the last 2 months
* Active substance abuse with alcohol or drugs
* Uncontrolled hypertension
* Liver disease
* Calcitonin level of ≥20 ng/L if eGFR ≥60 mL/min/1.73 m2 or ≥35 ng/L if eGFR <60 mL/min/1.73 m2
* Family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* History of active or untreated malignancy or are in remission from a clinically significant malignancy (other than basal- or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years
* Severe anemia
* Pregnant or breastfeeding
* Metal implants that preclude MRI testing
* Use of medications that are known to affect the study outcome measures
* Do not agree to use contraception throughout the study period in male and female participants of reproductive and childbearing age
* Persons who are not able to grant voluntary informed consent
* Unable or unwilling to follow the study protocol
* Have any other condition not listed in this section (e.g. hypersensitivity or intolerance) that is a contraindication of GLP-1R agonists

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Change in body weight | After 24 weeks of intervention
  Percent change in body weight
Change in body weight | After 52 weeks of intervention
  Percent change in body weight

SECONDARY OUTCOMES:
Proportion of participants losing at least 5% in body weight | After 24 weeks of intervention
  Proportion of participants in each group that lose at least 5% in body weight
Proportion of participants losing at least 5% in body weight | After 52 weeks of intervention
  Proportion of participants in each group that lose at least 5% in body weight
Proportion of participants losing at least 10% in body weight | After 24 weeks of intervention
  Proportion of participants in each group that lose at least 10% in body weight
Proportion of participants losing at least 10% in body weight | After 52 weeks of intervention
  Proportion of participants in each group that lose at least 10% in body weight
Proportion of participants losing at least 15% in body weight | After 24 weeks of intervention
  Proportion of participants in each group that lose at least 15% in body weight
Proportion of participants losing at least 15% in body weight | After 52 weeks of intervention
  Proportion of participants in each group that lose at least 15% in body weight
Fat mass and fat free mass | Before and after 24 weeks of intervention
  Fat mass and fat free mass will be assessed using dual-energy x-ray absorptiometry (DXA)
Fat mass and fat free mass | Before and after 52 weeks of intervention
  Fat mass and fat free mass will be assessed using dual-energy x-ray absorptiometry (DXA)
β-cell function | Before and after 24 weeks of intervention
  β-cell function will be assessed from a modified 3-hour oral glucose tolerance test
β-cell function | Before and after 52 weeks of intervention
  β-cell function will be assessed from a modified 3-hour oral glucose tolerance test
Insulin clearance | Before and after 24 weeks of intervention
  Insulin clearance will be assessed from a modified 3-hour oral glucose tolerance test
Insulin clearance | Before and after 52 weeks of intervention
  Insulin clearance will be assessed from a modified 3-hour oral glucose tolerance test
Plasma lipids | Before and after 24 weeks of intervention
  Fasting plasma lipid profile will be assessed by routine blood tests
Plasma lipids | Before and after 52 weeks of intervention
  Fasting plasma lipid profile will be assessed by routine blood tests
Blood pressure | Before and after 24 weeks of intervention
  Systolic and diastolic blood pressure will be measured
Blood pressure | Before and after 52 weeks of intervention
  Systolic and diastolic blood pressure will be measured
Sleep quality | Before and after 24 weeks of intervention
  Sleep quality will be assessed by polysomnography.
Sleep quality | Before and after 52 weeks of intervention
  Sleep quality will be assessed by polysomnography.
Sleep quantity | Before and after 24 weeks of intervention
  Sleep quantity will be assessed by polysomnography.
Sleep quantity | Before and after 52 weeks of intervention
  Sleep quantity will be assessed by polysomnography.
Liver fat | Before and after 24 weeks of intervention
  Liver fat will be assessed by using ultrasound
Liver fat | Before and after 52 weeks of intervention
  Liver fat will be assessed by using ultrasound
Intra-abdominal fat mass and intrahepatic triglyceride content | Before and after 52 weeks of intervention
  Intra-abdominal fat mass and intrahepatic triglyceride content will be assessed via magnetic resonance imaging (MRI)
Physical performance | Before and after 24 weeks of intervention
  Physical performance will be measured as the time in seconds that takes to walk 50 ft and to stand up 5 times from a chair.
Physical performance | Before and after 52 weeks of intervention
  Physical performance will be measured as the time in seconds that takes to walk 50 ft and to stand up 5 times from a chair.
Grip strength | Before and after 24 weeks of intervention
  Grip strength will be measured using a hand dynamometer.
Grip strength | Before and after 52 weeks of intervention
  Grip strength will be measured using a hand dynamometer.
Lifestyle program adherence | After 24 weeks of intervention
  Number of sessions attended
Lifestyle program adherence | After 52 weeks of intervention
  Number of sessions attended
Drug/placebo adherence | After 24 weeks of intervention
  Number of injections received
Drug/placebo adherence | After 52 weeks of intervention
  Number of injections received
Program acceptability from community health workers and study participants | After 24 weeks of intervention
  Community health workers' and study participants' perceptions of program acceptability via questionnaire
Program acceptability from community health workers and study participants | After 52 weeks of intervention
  Community health workers' and study participants' perceptions of program acceptability via questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Jacome Sosa, Principal Investigator — Washington University School of Medicine
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States